CLINICAL TRIAL: NCT07200453
Title: Development and Effectiveness Evaluation of an Interactive E-learning Environment to Enhance Digital Health Literacy in Cancer Patients: Study Protocol for a Randomized Controlled Trial
Brief Title: Evaluation of an Interactive E-learning Environment to Enhance Digital Health Literacy in Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: German Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: S-158/2024
Record Dates: First submitted 2024-07-30; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Neoplasms
Keywords: digital health; eHealth; health literacy; eHealth literacy; health information; e-learning; medical education; digital health literacy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This trial is designed as a randomized controlled superiority trial with five parallel groups and a primary endpoint of digital health literacy. The study also includes intervention development and pre-testing. Randomization will be performed as a proportionally stratified randomization with variable block length and 1:1:1:1:1 allocation.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding will be maintained throughout the duration of the study to increase the objectivity of the results and to minimize the influence of participants' expectations on the study results. Participants in the control group will not receive any intervention and will be referred to the CIS brochure "Your journey through cancer", which will not include any information on how to search for cancer-related information online. In the dataset and in REDCap, the 5 randomization groups are referred to as groups A, B, C, D and E, so that it is not clear to the research staff evaluating the data which intervention the patients received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- e-learning - intervention group 1.1 (Experimental): Participants in intervention group 1.1 will be given access to an e-learning environment with all the persuasive primary task support elements (reduction, tunneling, rehearsal). Participants can complete the e-learning within 2 weeks. The e-learning program takes approximately 20-45 minutes to complete.
  Interventions: Behavioral: intervention group 1.1 - e-learning
- e-learning - intervention-group 1.2 (Experimental): Participants in intervention group 1.2 are given access to the same e-learning environment without the persuasive primary task support element, tunneling. Tunneling means that the educational content is organized step by step in separate chapters of the program. Participants can complete the e-learning within 2 weeks. The e-learning program takes approximately 20-45 minutes to complete.
  Interventions: Behavioral: intervention-group 1.2 - e-learning
- e-learning - intervention-group 1.3 (Experimental): Participants in intervention group 1.3 are given access to the same e-learning environment without the persuasive primary task support element, rehearsal. All rehearsal elements such as quizzes will be removed from the e-learning environment. Participants can complete the e-learning within 2 weeks. The e-learning program takes approximately 20-45 minutes to complete.
  Interventions: Behavioral: intervention-group 1.3 - e-learning
- PDF document - intervention-group 2 (Active Comparator): This intervention group is given access to a PDF document with the same content as in the e-learning environment. Participants can complete the website content within 2 weeks. The PDF document takes approximately 20-45 minutes to complete.
  Interventions: Behavioral: intervention-group 2 - PDF
- No Intervention/ treatment as usual (No Intervention): The last group (treatment as usual) receives no intervention. However, they are sent a brochure that has nothing to do with digital health literacy.

INTERVENTIONS:
Behavioral: intervention group 1.1 - e-learning — The e-learning environment will include text, images, and short videos created using Articulate Rise 360, an easy-to-use e-learning authoring tool, with the following content to improve the different skills of digital health literacy:
  1. Evaluating reliability skills: Participants will get to know criteria and indicators for evaluating the content of the information they find and for assessing the trustworthiness of website providers.
  2. Improving information skills: Participants will learn simple rules on how to optimize their Google searches.
  3. Improving navigation skills: Participants will learn simple rules for navigation; using the back button; using more than one tab; drop-down lists and anchor links are introduced.
  4. Additional goals are to raise awareness about various aspects related to online searches, including the exploration of alternative and complementary therapies, and the importance of data protection.
  Arms: e-learning - intervention group 1.1
Behavioral: intervention-group 1.2 - e-learning — Participants are also given access to the e-learning environment. However, they will not be taken step-by-step through the content (tunneling). They can choose the order of the content.
  Arms: e-learning - intervention-group 1.2
Behavioral: intervention-group 1.3 - e-learning — Participants are also given access to the e-learning environment, but all rehearsal elements such as quizzes will be removed from the e-learning environment.
  Arms: e-learning - intervention-group 1.3
Behavioral: intervention-group 2 - PDF — Participants in IG2 will receive the same content as participants in the IG1.1, but not within the interactive learning environment, but in a non-interactive PDF format.
  Arms: PDF document - intervention-group 2

SUMMARY:
This study aims to create and test an online learning tool to help people with cancer improve their skills in finding and understanding health information online. The main question it aims to answer is:

• Do people with cancer who use the online learning tool improve their skills more than those who don't use the tool?

The investigators will test this idea in a study. The investigators will put people into different groups by chance and compare the results. 660 people with cancer will participate. These people will be chosen to represent different types of cancer.

* Group 1: Uses the online learning too (3 versions)
* Group 2: Uses a PDF with the same information
* Control Group: Receives no intervention

What Participants Will Do:

Use the online tool or PDF to learn how to find reliable cancer information online.

Answer questions about their digital health skills before starting, after 2 weeks, and after 8 weeks.

Development:

Before the start of the main study the online tool will be developed and tested. The investigators will first show a prototype of the tool to two discussion groups and use their feedback to improve it. Then, experts and people with cancer will test the final version

DETAILED DESCRIPTION:
Background: The Internet allows cancer patients to access information about their disease at any time. However, the quality of online information varies widely. Information is often inaccurate or does not provide all the details patients need to make informed decisions. Patients' often inadequate ability to find and critically evaluate cancer-related information online can lead to misinformation.

Objective: An interactive e-learning environment to promote digital health literacy will be developed and evaluated for effectiveness. The primary hypothesis is: Cancer patients who use the e-learning environment (IG1.1-IG1.3) or the content of the environment as a non-interactive PDF file (IG2) will show greater improvement in their digital health literacy from baseline to eight weeks after baseline compared to patients who do not receive such an intervention.

Methods: The hypothesis will be tested in a randomized controlled trial (RCT). In the e-learning environment, patients will learn strategies (e.g., checking information on different websites) to use when searching for reliable cancer-related online information. During the development, a prototype will be presented to two focus groups. The results of the focus groups will be implemented in a final prototype. The usability of this prototype will then be tested by usability experts and patients. 660 cancer patients will be recruited and randomly assigned in a 3:1:1 ratio to IG1.1-IG1.3 (three variants of the environment), IG2 (a PDF containing the same content as the environment), or the control group. Two thirds of the 660 participants will be recruited through the German Cancer Information Service (CIS) and one third will be recruited through non-CIS routes. A proportionally stratified sample will be drawn according to the cancer incidence. The primary outcome, digital health literacy, will be measured at baseline, two weeks, and eight weeks after baseline.

ELIGIBILITY:
Inclusion criteria:

* cancer diagnosis
* sufficient knowledge of the German language as all study content and questionnaires will be in German only
* Participants must also have and be able to use a digital device (smartphone, tablet, PC, laptop, etc.) with an internet connection
* Confirm consent to participate in the study

Exclusion criteria:

* Patients who are severely cognitively impaired due to their cancer or other illness
* Patients who are unable to operate a digital device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the patient-reported digital health literacy measured by the Digital health literacy Instrument (DHLI) at 8 weeks | The questionnaire will be administered at baseline (TO), follow-up at 2 weeks (T1), and follow-up at 8 weeks (T8).
  The primary outcome is the patient-reported digital health literacy based on the German version of the Digital health literacy Instrument (DHLI), resulting from the mean of the 21 items included. All 21 items are answered on a four-point scale (1="very difficult" to 4="very easy" and from 1="never" to 4="often"). A higher mean score indicates higher digital health literacy.

SECONDARY OUTCOMES:
Digital health literacy measured with the performance-based items of the DHLI | The questionnaire will be administered at baseline (TO), follow-up at 2 weeks (T1), and follow-up at 8 weeks (T8).
  The digital health literacy of the participants will also be measured using six performance-based items of the DHLI - one item each for the sub-skills: operational skills, navigation skills, evaluating reliability, information searching, determining relevance and protecting privacy. Responses will be coded as correct (score=1) or incorrect (score=0) and then the scores of all six items will be added together to form a total score.
Participants' motivation to use the e-learning environment measured with the Reduced Instructional Materials Motivation (RIMMS) | The questionnaire will be administered at follow-up at 2 weeks (T1).
  The RIMMS is a 4-dimensional (attention, relevance, confidence, satisfaction), 12-item short version of the "Instructional Materials Motivation Survey". The items will be rated by the participants on a 5-point scale from 1="strongly disagree" to 5="strongly agree". The resulting mean value across all 12 items will be used for the overall assessment of motivation.
Acceptability of the e-learning environment as measured by the Acceptability of Intervention Measure (AIM) questionnaire. | The questionnaire will be administered at follow-up at 2 weeks (T1).
  The AIM contains 4 items that will be rated by the participants on a 5-point scale from 1 = "disagree" to 5 = "agree". Acceptability will be reported as the mean value of the four items, with a higher score indicating greater acceptance.
Appropriateness of the e-learning environment as measured by the Intervention Appropriateness Measure (IAM) questionnaire. | The questionnaire will be administered at follow-up at 2 weeks (T1).
  The IAM contains 4 items that will be rated by the participants on a 5-point scale from 1 = "disagree" to 5 = "agree". Appropriateness is presented as the mean value of the four items, with a higher score indicating greater appropriateness.
Feasibility of the e-learning environment as measured by the Feasibility of Intervention Measure (FIM) questionnaire. | The questionnaire will be administered at follow-up at 2 weeks (T1).
  The FIM contains 4 items that will be rated by the participants a 5-point scale from 1 = "disagree" to 5 = "agree". Feasibility is presented as the mean value of the four items, with a higher score indicating greater feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Holger Schulz, Prof., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf; Susanne Weg-Remers, Dr., Principal Investigator — German Cancer Research Center
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
* The study protocol was submitted to Frontiers in Public Health on June 24, 2024.
  * The statistical analysis plan will be uploaded prior to unblinding for data analysis.
  * The study data will be made available to other scientists via the online open access repository Figshare (https://figshare.com/) Figshare uses Creative Commons licenses, which give other researchers the right to use and build upon a dataset.
Supporting Information: SAP
Time Frame: The data will be available a few days before the study results are released.
Access Criteria: Figshare uses Creative Commons licenses, which give other researchers the right to use and build upon a dataset.

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-08-28): https://cdn.clinicaltrials.gov/large-docs/53/NCT07200453/SAP_000.pdf